CLINICAL TRIAL: NCT00236496
Title: A Comparison of the Efficacy and Safety of Topiramate Versus Placebo in the Treatment of Essential Tremor
Brief Title: A Comparison of the Efficacy and Safety of Topiramate Versus Placebo in Treating Tremor of Unknown Cause.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002659
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Essential Tremor
Keywords: tremor; essential tremor
MeSH Terms: conditions — Essential Tremor; Tremor | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of topiramate as compared to placebo in treating patients with tremor of unknown cause.

DETAILED DESCRIPTION:
Essential tremor is a very common form of tremor, occurring in up to 5% of people. It may be inherited. In 90% of patients, the tremor is in the hands; however, it can also be in the head, voice, legs, jaw, and tongue. Essential tremor may be treated by the blood pressure medicine propranolol or the anti-seizure drug primidone. The drawbacks of these drugs are that they tend to lose effectiveness over time, and they may cause side effects. Researchers believe that topiramate, an anti-seizure drug, may be effective in treating essential tremor. In this double blind, placebo-controlled study, patients with essential tremor will start at a low dose of topiramate (25 milligrams) or placebo. The dose will be gradually increased over 12 weeks to a maximum of 400 milligrams daily, taken in two divided doses. Then, each patient will stay on the established dose for the next 12 weeks. During the next phase of the study, the patients will slowly reduce the dose until they stop taking the study drug, after which, patients have the option of taking up to 600 milligrams of topiramate (not placebo) in a 14-week extension of the study. This study was designed to investigate the hypothesis that topiramate will be more effective than placebo in the treatment of essential tremor as measured by the Clinical Rating Scale for Tremor (TRS) and is well tolerated. The TRS is a three part scale that measures tremor location/severity rating, specific motor tasks/function rating, and functional disabilities resulting from tremor. Safety evaluations are assessed throughout the study.

Topiramate or placebo, starting with a dose of 25 mg, then gradually increased over 12 weeks up to 400 mg daily (two 100-mg tablets taken by mouth twice a day) and continued on this dose for 12 weeks in the maintenance phase; up to 600 milligrams of topiramate in the open-label phase.

ELIGIBILITY:
Inclusion Criteria:

* Current symptoms of essential tremor based on the Tremor Investigational Group (TRIG) criteria
* Dominant upper extremity posture or action intention tremor of 2 (moderate) to 4 (severe)
* In good health otherwise

Exclusion Criteria:

* Patients with abnormal neurologic signs other than essential tremor
* Taking more than one anti-tremor medication
* Taking drugs known to cause tremors
* With physical damage to the nervous system or Parkinson's disease
* Known to be abusing drugs or alcohol
* Women who are pregnant or breast-feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2001-10; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Clinical Rating Scale for Tremor (TRS) score at Visit 8 (or patient's final visit) of the double-blind phase

SECONDARY OUTCOMES:
TRS subscale scores; composite normalized score; overall TRS score; patient and investigator assessment scores.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Comparison of the Efficacy and Safety of Topiramate Versus Placebo in the Treatment of Essential Tremor — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=485&filename=CR002659_CSR.pdf